CLINICAL TRIAL: NCT00383877
Title: Effect of Insulin Detemir on Blood Glucose Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1684
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH

SUMMARY:
This trial is conducted in China. This trial aims for a comparison of the effect on glycemic control in subjects with type 2 diabetes of insulin detemir or NPH-insulin given once daily at bedtime as add-on to oral anti-diabetic drug(s).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1C greater than 7.5% and less than or equal to 11.0%
* Currently on any oral antidiabetic drug (OAD) more than or equal to 3 months

Exclusion Criteria:

* Previous acute treatment with insulin for more than 7 days.
* Treatment with OAD(s) which does not adhere to the approval labeling.
* Proliferate retinopathy or maculopathy that has required acute treatment within the last year.
* Known hypoglycaemia unawareness or recurrent major hypoglycaemia, that may interfere with study participation as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 20 weeks of treatment

SECONDARY OUTCOMES:
FBG | after 20 weeks of treatment
Safety profile | during 20 weeks treatment
Proportion of subjects achieving HbA1c less than or equal to 7.0% | after 20 weeks of treatment
Within-subject variation of self measured blood glucose (SMBG) before breakfast during the trial at the end of the trial | before breakfast during the trial at the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com